CLINICAL TRIAL: NCT01083563
Title: The Morphologic and Functional Relationship Between the Draining PLN and Synovial Inflammation in the Knee Joints of RA Patients Before and After Anti-TNF or B Cell Depletion Therapy
Brief Title: Draining PLN and Synovial Inflammation in RA Knee Joints Pre and Post Anti-TNF or B Cell Depletion Therapy
Status: Terminated | Type: Observational
Why Stopped: Funding has ended prior to complete enrollment
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Christopher Ritchlin, M.D., M.P.H., Professor of Medicine Allergy, Immunology & Rheumatology Division, University of Rochester
Other Study IDs: RSRB-27325
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Rheumatoid Arthritis
Keywords: TNF; CD20; RA
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RA inadequate response to methotrexate: Individuals with rheumatoid arthritis who have had an inadequate response to methotrexate and will be starting on an anti-TNF agent.
- RA inadequate response to anti-TNF.: Individuals with rheumatoid arthritis who have had an inadequate response to an anti-TNF and will be be given a rituximab infusion.

SUMMARY:
The purpose of this study is to examine the effect of anti-TNF therapy on rheumatoid arthritis using magnetic resonance imaging (MRI) and ultrasound imaging.

Anti-TNF therapies include a group of medications such as Enbrel, Remicade and Humira that affect your body's inflammatory response. These medications are routinely prescribed for the treatment of rheumatoid arthritis.

DETAILED DESCRIPTION:
The specific aim of this study is to examine the morphologic and functional relationship between the draining PLN and synovial inflammation in the knee joints of RA patients before and after therapy with TNF antagonists or B cell depletion therapy. The extensive search for informative and practical clinical biomarkers of RA has produced several candidates including CRP, anti-CCP antibodies and matrix metalloproteinase-3 (MMP-3), but none of these soluble molecules can predict disease progression with a high degree of certainty, and no biomarker has been identified that can predict flare. Thus, our findings that PLN collapse precedes arthritis flare in the murine model offers a novel biomarker that may be of great value in RA, but requires validation in humans. To this end, we propose two clinical pilots that are designed to test the validity and feasibility of PLN assessment and quantification in active RA by 3T CE-MRI and Doppler US. The second goal of these pilots is to see if there is a relationship between the clinical response to either a TNF antagonist or B cell depletion and a change in the size or CE pattern of PLN. The pilot studies outlined below are designed to test the hypotheses that an effective clinical response to anti-TNF or BCDT is associated with an increase in draining LN function. While our overall goal is to determine if Doppler US can predict flare, we must first establish the validity and feasibility of this approach so that we can design a clinical trial that is properly designed and adequately powered.

Aim A: To assess the effect of TNF inhibition on volume and CE in the PLN in RA patients by MRI, and compare the effectiveness of Doppler US to achieve the same outcome measures.

Hypothesis: Rheumatoid synovitis in the knee is triggered by TNF over-expression by monocytes/macrophages in the synovium and/or the draining PLN, which produces inflammation that exceeds PLN draining capacity. This results in decreased inflammatory cell egress from the joint and arthritic flare. Effective anti-TNF therapy in RA will result in increased PLN function due to decreased cellularity and lymphatic flow from the synovium to the draining node.

Rationale: To address our first hypothesis, we plan to determine the validity and feasibility of draining LN function by analyzing the ability of 3T CE-MRI and Doppler US to quantify PLN in inflamed RA knees. While CE-MRI (volume x CE) will be the primary outcome measure of PLN function based on our pre-clinical studies, this approach is not adaptable to standard clinical practice. Furthermore, serial MRIs to monitor flare in RA are not feasible due to cost, time, convenience and availability of resources. Thus, parallel US studies will be performed to determine if this instrument, which is gaining acceptance in rheumatology practice, can generate accurate and quantifiable PLN measurements.

Aim B. To assess the effect of anti-CD20 therapy on volume and CE in the PLN in RA patients who "flare" after a period of effective anti-TNF therapy.

Hypothesis: RA flare in patients who had been effectively managed by anti-TNF therapy is caused by a local insult that triggers B-cell migration and precipitates LN shutdown and decreased inflammatory cell egress from the joint. Effective anti-CD20 BCDT therapy in these patients will correlate with increased PLN function and decreased inflammation in the synovium.

Rationale: RA is a complex syndrome in which excess TNF production is central to disease pathogenesis. While ~70% of these patients can be effectively managed by anti-TNF therapy, an additional insult (i.e. local immune response or trauma) results in a flare that cannot be adequately suppressed by standard anti-TNF therapy in some patients (80, 81). Many patients who flare on one or more anti-TNF therapies do respond to BCDT (26). An explanation for this that fits our preliminary findings in the TNF-Tg mice is that a local immune-inflammatory response that shares lymphatics with RA synovium can induce CXCL13 expression in monocyte/macrophages in the draining LN and these cells and soluble CXCL13 enter the LN via the lymphatics and triggers mass migration of B-cells into the paracortical sinuses. This B cell translocation results in decreased egress of inflammatory cells, which had been maintained by anti-TNF therapy, and manifests as an arthritic flare. To provide a human correlate for the murine experiments designed to test this hypothesis outlined in Aim 2, and to produce feasibility data for a clinical trial to test this novel mechanism of action, we will evaluate PLN radiographic changes following anti-CD20 BCDT in RA patients who flare on anti-TNF therapy. We will also assess DAS28 clinical responses.

ELIGIBILITY:
Inclusion Criteria

* Signed, IRB-approved, written informed consent
* Subjects can be of either gender but must be more than 18 years old.
* Subjects must fulfill the disease activity criteria for RA and a DAS28 will be assessed at baseline and at 2 months after rituximab therapy.
* Aim A - Eligible subjects must meet criteria for RA and have an inadequate response to MTX defined as DAS28 >5.1. They must have been on a steady dose of MTX (between 15 and 20 mg /week for a minimum of 8 weeks). Subjects must have evidence of knee synovitis on exam to enter the study.
* Aim B - Subjects must have demonstrated a response to a TNF antagonist as evidenced by a DAS score <2.8 or <4 tender and swollen joints. Flare will be defined as a DAS 28 >5.1 of more than 8 swollen and tender joints. Subjects must have evidence of knee synovitis to enter the study. Subjects will be off etanercept, infliximab or adalimumab for 4 weeks before starting BCDT. All subjects must also be on a stable dose of DMARD (MTX, leflunomide, azulfidine, hydroxychloroquine) for 8 weeks before entry into the study.

Exclusion Criteria

* Patients will be excluded for medical or other reasons at the discretion of the investigators. The reasons for the exclusion must be recorded, e.g. risk of non-compliance, vulnerability, medically unstable, etc.
* Active systemic disorders or inflammatory conditions (i.e., chronic infection with hepatitis B, hepatitis C or HIV) other than the conditions being studied.
* Patients with a plasma creatinine > 1.5 mg/dl
* Aim B - Subjects with an allergy to corticosteroids will be excluded from the study.
* Anyone answering yes to the following questions will be excluded:

Do you have a history of:

1. Cardiac (Heart) pacemaker or defibrillator?
2. Cardiac (Heart) valve replacement or prosthesis?
3. Aneurysm clips from brain surgery?
4. Ear prosthesis (cochlear or stapedial implant)? (hearing aids?)
5. Neurostimulator?
6. Biostimulator?
7. Any type of pumps in or on your body?
8. Shrapnel, gunshot wound, BB pellet?
9. Metallic penile prosthesis?
10. Metallic blood vessel filter or stent?
11. Orthopedic prosthesis?
12. Have you ever had an injury involving metal fragments in your eye?
13. Have you ever had neurosurgery (brain or skull surgery)?

Note: Subjects treated with rituximab will not be excluded from study based on their immunosuppressive drugs but use of these agents will be recorded and discussed in the analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female RA sufferers not less than 18 yrs of age who are currently experiencing knee synovitis. Racial and ethnic origin of subjects will be monitored to reflect the diversity of our community.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2009-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Morphologic and functional relationship between the draining PLN and synovial inflammation in the knee joints of RA patients | Week 0 (initial medication dose) and Week 8 (post medication dose)
  To examine the morphologic and functional relationship between the draining PLN and synovial inflammation in the knee joints of RA patients before and after therapy with TNF antagonists or B cell depletion therapy via MRI and Doppler ultrasound.
TNF inhibition on volume and CE in the PLN in RA patients by MRI versus Doppler ultrasound. | Week 0 (initial medication dose) and Week 8 (post medication dose)
  To assess the effect of TNF inhibition on volume and CE in the PLN in RA patients by MRI, and compare the effectiveness of Doppler US to achieve the same outcome measures.
Effect of anti-CD20 therapy on volume and CE in the PLN in RA patients who "flare" | Week 0 (initial medication dose) and Week 8 (post medication dose)
  To assess the effect of anti-CD20 therapy on volume and CE in the PLN in RA patients who are experiencing knee synovitis after a period of effective anti-TNF therapy

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ritchlin, MD / MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Rahimi H, Bell R, Bouta EM, Wood RW, Xing L, Ritchlin CT, Schwarz EM. Lymphatic imaging to assess rheumatoid flare: mechanistic insights and biomarker potential. Arthritis Res Ther. 2016 Sep 1;18:194. doi: 10.1186/s13075-016-1092-0. PMID 27586634
- [Derived] Li J, Zhou Q, Wood RW, Kuzin I, Bottaro A, Ritchlin CT, Xing L, Schwarz EM. CD23(+)/CD21(hi) B-cell translocation and ipsilateral lymph node collapse is associated with asymmetric arthritic flare in TNF-Tg mice. Arthritis Res Ther. 2011 Aug 31;13(4):R138. doi: 10.1186/ar3452. PMID 21884592